CLINICAL TRIAL: NCT00506883
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group, 1 Week, Dose Comparison Study to Evaluate the Efficacy, Safety, and Tolerability of MPC-004 in Patients With an Acute Gout Flare
Brief Title: MPC-004 for the Treatment of an Acute Gout Flare
Acronym: AGREE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Matthew Davis, MD, AR Scientific
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPC 004-06-3001
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Colchicine (Experimental): After confirmation of a gout flare, patients were to begin standard dosing of colchicine 4.8mg (two capsules (1.8mg) initially followed by additional one capsule doses (0.6mg) every hour for an additional 6 doses).
  Interventions: Drug: High Dose Colchicine (4.8 mg total dose)
- Low Dose Colchicine (Experimental): Within 12 hours of a confirmed gout flare, patients were to begin the low dose colchicine regimen consisting of a total dose of 1.8 mg - two colchicine capsules initially (1.2 mg)followed an hour later by a single additional capsule of active drug(0.6 mg)then by 5 additional hourly doses of an identical looking placebo capsules
  Interventions: Drug: Low Dose Colchicine (1.8mg total dose)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: High Dose Colchicine (4.8 mg total dose) — At randomization, patients were given an identical looking blister pack containing (8) over encapsulated colchicine 0.6 mg tablets identical in appearance to placebo capsules. Patients were instructed to take 2 capsules initially (1.2 mg) followed by an additional capsule (0.6 mg) every hour for a total of six additional doses (total colchicine dose 4.8 mg) beginning within 12 hours of onset of a qualifying gout flare as confirmed by calling the gout flare call center.
  Other Names: Colcrys TM, Colchicine 0.6 mg
  Arms: High Dose Colchicine
Drug: Low Dose Colchicine (1.8mg total dose) — At randomization, patients were given an identical looking blister pack containing (3) over encapsulated colchicine 0.6 mg tablets identical in appearance to placebo capsules and five placebo capsules. Patients were instructed to take 2 capsules initially (0.6 mg x 2) followed by an additional capsule every hour for a total of six additional doses (one active (0.6 mg) and 5 placebo capsules), a total colchicine dose = 1.8 mg) beginning within 12 hours of onset of a qualifying gout flare as confirmed by calling the gout flare call center
  Other Names: Colcrys TM, Colchicine 0.6 mg
  Arms: Low Dose Colchicine
Other: Placebo Control — At randomization, patients were given an identical looking blister pack containing (8) placebo capsules identical in appearance to the study drug. Patients were instructed to take 2 capsules initially followed by an additional capsule every hour for a total of six additional doses beginning within 12 hours of onset of a qualifying gout flare as confirmed by calling the gout flare call center.
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel group, dose-comparison to determine the efficacy and safety of a standard-dose of colchicine (4.8 mg) versus low-dose colchicine (1.8 mg) or placebo for acute gout flares.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, double-blind, placebo-controlled, parallel group trial to compare the efficacy and safety of standard-dose colchicine (STD)(total dose = 4.8 mg) versus low-dose colchicine (total dose 1.8 mg) or placebo for the treatment of acute gout flares. Eight hundred and thirteen patients with a confirmed diagnosis of gout were screened. 238 of the screened patients failed screening; 235(98.7%) failed because they did not meet inclusion/exclusion criteria. The 575 eligible patients were randomly assigned (1:1:1) to one of three treatment groups . At the randomization visit the investigator dispensed a blister card containing eight identical looking capsules (in a combination of active drug and placebo capsules) in a double blind fashion for use during their next gout flare. Patients were instructed to self-initiate treatment with the study medication within 12 hours of a gout flare onset. Gout flares were determined by calling a Gout Flare Call Center established for this purpose. At Investigator discretion, rescue medication could also be provided, but patients were encouraged not to use rescue medication within the first 24 hours after starting treatment with study drug. Of the 575 study participants, 185 had a qualifying gout flare and 390 did not. Patients used a diary to record study drug administration, pain score, the presence or absence of gastrointestinal adverse events (nausea, vomiting, diarrhea, and abdominal pain) and the timing of any rescue medication use prior to beginning treatment and 1, 2, 3, 4, 5, 6, 7, 8, 16, 24, 32, 40, 48, 56, 64, and 72 hours after the start of dosing.

The pain score was based on a scale of 1 - 10 where 1 was no pain and 10 was the worst pain imaginable. Efficacy was defined as a 50% reduction in pain score in the target joint at 24 hours in patients who did not use rescue medicine. The primary efficacy analysis was to be based on an Intent-to-Treat (ITT) population, defined as all patients who were randomized, contacted the Call Center, and were instructed to begin taking study drug. An otherwise qualified patient was excluded from the ITT population only if the patient returned a study drug blister pack completely unused.

Secondary outcome measures compared the efficacy of STD dose colchicine to a low dose regimen and placebo using the same criteria for efficacy as for the primary outcome measure.

Additional secondary outcome measures were time to 50% and 90% reduction in pain in the target joint analyzed by treatment group using Kaplan-Meier methods, and the change in mean pain intensity from 0 to 72 hours plotted by time point for each treatment group.

All safety analyses were carried out using the safety population defined as all patients who received at least one dose of study medication regardless of authorization by the Call Center To determine the safety of colchicine when administered via two different dose regimens all patients who had a gout flare were seen by the investigator as soon as possible after onset and evaluated until the flare and any adverse events resolved. All adverse effects, whether recorded by the patient in the diary or obtained by systematic evaluation by the investigator were recorded and reported in tabular form. Treatment-emergent adverse events (TEAE) were summarized by MedDRA System Organ Class and preferred terms and tabulated according treatment arm, overall incidence, severity and relationship to study medication. Multiple events within a patient were counted once and at greatest severity and closest relationship to study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender and of any race ≥18 years of age.
2. If female, patients must be postmenopausal as evidenced by lack of menses for ≥12 consecutive months.
3. Patients must present with a confirmed diagnosis of gout.
4. Patients must have experienced ≥2 acute gouty arthritic attacks in the 12 months prior to randomization.
5. Patients on urate lowering therapy must be on a stable dose and schedule with no changes in therapy for 4 weeks prior to randomization and expected to remain on a stable regimen during study participation.
6. Patients must be willing to adhere to the study schedule and the protocol requirements.
7. Patients must be willing and able to give written informed consent. A HIPAA and/or state privacy consent must also be signed.

Exclusion Criteria:

1. Patients with acute polyarticular gout (>4 joints).
2. Patients who have experienced >2 acute gouty arthritic attacks per month, or >12 attacks overall, in the 6 months prior to randomization.
3. Patients with arthritis due to any cause other than gout that may confound any study assessments per Investigator discretion.
4. Patients with a history of myocardial infarction, unstable angina, cerebrovascular events, or coronary artery bypass grafting within the previous 6 months prior to screening.
5. Patients with active myeloid leukemia, obstructive gastrointestinal cancer, or metastatic cancer.
6. Patients with chronic renal dysfunction (creatinine clearance <60 mL/min as estimated with the Cockcroft Gault formula).
7. Patients with chronic hepatic dysfunction.
8. Patients with a history of alcohol or substance abuse within the 12 months prior to randomization.
9. Patients who have any concomitant illness or other finding that, in the opinion of the Investigator, would confound the study data or place the patient at unacceptable risk if the patient were to participate in the study, or that would require frequent adjustments in concomitant medications during the course of the study.
10. Patients using systemic corticosteroid, cyclosporine, adalimumab, etanercept, infliximab, anakinra, abatacept, mycophenolate, azathioprine, anticoagulants (warfarin, heparin, low molecular weight heparin [LMWH], antithrombin agents, thrombin inhibitors, or selective Factor Xa inhibitors [note, use of aspirin ≤325 mg/day is allowed]), or chronic use of non steroidal anti inflammatory drugs (NSAIDs), acetaminophen, tramadol, and other analgesics such as opiates at screening
11. Use of any investigational drug within 30 days prior to randomization.
12. Patients currently participating in another research study or anticipated to enroll in such during participation in this study.
13. Patients for whom informed consent cannot be obtained.
14. Patients who have previously been randomized into this study and begun ingestion of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Davis, MD, RPh, Study Chair — AR Scientific, Inc.
Locations (83):
- United States (83):
  - Innovative Clinical Trials, Birmingham, Alabama
  - Birmingham, Alabama
  - Tomac, Inc., Columbiana, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Genova Clinical Research, Tucson, Arizona
  - Tucson, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Irvine Center for Clinical Research, Irvine, California
  - La Jolla, California
  - Paramount, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - San Diego, California
  - West Covina, California
  - Florida Medical Center, Clearwater, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - George E. Platt, MD, Green Cove Springs, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Lake Mary, Florida
  - Medical Research Trust, Lake Worth, Florida
  - Hillcrest Medical Center, Orange City, Florida
  - Farmer MD, PA, Ormond Beach, Florida
  - Coastal Medical Research, Inc., Port Orange, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Geodessey Research, LLC, Vero Beach, Florida
  - Bond Clinic, Winter Haven, Florida
  - Global Research Partners & Consultants, Inc., Calhoun, Georgia
  - Decatur, Georgia
  - North Georgia Rheumatology Group, PC, Lawrenceville, Georgia
  - Arthritis & Osteoporosis Center of South Georgia, Tifton, Georgia
  - Boise, Idaho
  - Idaho Arthritis & Osteoporosis Center, Meridian, Idaho
  - Lake County Research Associates, Libertyville, Illinois
  - Moline, Illinois
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - The Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - David H. Neustadt PSCq, Louisville, Kentucky
  - Gulf Coast Research, Baton Rouge, Louisiana
  - Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - Rockville, Maryland
  - The Center for Rheumatology & Bone Research, Wheaton, Maryland
  - Future Care Studies, Springfield, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Justus Fiechtner, MD, MPH, Lansing, Michigan
  - Arthritis Associates, Hattiesburg, Mississippi
  - Medical Center Healthcare Research, Florissant, Missouri
  - Medex Healthcare, St Louis, Missouri
  - Las Vegas, Nevada
  - Arthritis Center of Reno, Reno, Nevada
  - Arthritis & Osteoporisis Associates, Manalapan, New Jersey
  - Rheumatology and Arthritis Associates, Medford, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - Southwest Medical Associates, Brewster, New York
  - Concorde medical Group, New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Williamsville, New York
  - Arthritis Consultants of the Carolinas, Belmont, North Carolina
  - Arthritis & Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Dayton, Ohio
  - Mayfield Village, Ohio
  - Middleburg Heights, Ohio
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Orangeburg, South Carolina
  - Milan, Tennessee
  - New Tazewell, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Sugarland, Texas
  - Ettrick, Virginia
  - Portsmouth, Virginia
  - Reston, Virginia
  - Suffolk, Virginia

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Bennett K, Kook KA, Crockett RS, Davis MW. High versus low dosing of oral colchicine for early acute gout flare: Twenty-four-hour outcome of the first multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-comparison colchicine study. Arthritis Rheum. 2010 Apr;62(4):1060-8. doi: 10.1002/art.27327. PMID 20131255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 2007 between 4 April and 3 December 813 patients were screened at 74 US treatment centers. 72 centers randomized a total 575 patients. 185 patients at 54 centers had a qualifying gout flare and 184 are included in the ITT population. The remaining, 390 patients had no flare or had a flare that failed to qualify for study medication use
Pre-assignment Details: 813 patients with confirmed diagnosis of gout based on American College of Rheumatology criteria were screened. 575 patients qualified and were randomized within 28 days of screening. 238 patients failed screening. The vast majority, 235 (98.7%) failed to meet inclusion/exclusion criteria.
Groups:
- High Dose Colchicine(MPC-004): Standard Dose Colchicine - 4.8 mg (total dose): 1.2 mg of oral colchicine (2 x 0.6 mg tablets) at onset of confirmed gout flare followed by 0.6 mg oral colchicine (1 x 0.6 mg tablet) every hour for 6 hours. All doses were over encapsulated to mimic the appearance of the placebo.
- Low Dose Colchicine(MPC-004): Low Dose Colchicine - 1.8 mg (total dose): 1.2 mg of oral colchicine (2 x 0.6 mg tablets) at onset of confirmed gout flare followed by 0.6 mg oral colchicine (1 x 0.6 mg tablet) after 1 hours followed by placebo every hour thereafter hourly for 5 additional hours. All active doses were over encapsulated to mimic the appearance of the placebo.
- Placebo: Two oral placebo capsules at onset of a confirmed gout flare followed by 1 oral placebo capsule every hour for an additional 6 hours.
Period: Overall Study
Arm/Group | High Dose Colchicine(MPC-004) | Low Dose Colchicine(MPC-004) | Placebo
Started | 52 | 74 | 59
Completed | 45 | 71 | 55
Not Completed | 7 | 3 | 4
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Other | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Colchicine(MPC-004) | Low Dose Colchicine(MPC-004) | Placebo | Total
Number analyzed (Participants) | 52 | 74 | 59 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 61 | 53 | 160
  >=65 years | 6 | 13 | 6 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 51.9 (10.02) | 51.4 (11.79) | 51.2 (11.36) | 51.5 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 49 | 72 | 55 | 176

OUTCOME MEASURES:

1. Primary Outcome: Responders
Description: Responders were defined as patients who achieved a ≥ 50% reduction in target joint pain score from baseline at 24 hours without using rescue drug, using an 11 point scale from 0 to 10, with 10 being the worst pain imaginable after beginning therapy.
Time Frame: 24 hours after baseline
Population: The Intent-to-Treat (ITT) population(N=184) was used. The ITT group is defined as all patients who were randomized,and had a qualifying gout flare based on contact with the Gout Flare Call Center, who were instructed to begin taking and took at least one dose of the study drug study drug. One patient had a flare, but
Measure: Number; unit: Participants
Arm/Group | High Dose Colchicine(MPC-004) | Low Dose Colchicine(MPC-004) | Placebo
Number analyzed (Participants) | 52 | 74 | 58
Participants | 17 | 28 | 9

ADVERSE EVENTS:
Arm/Group | High Dose Colchicine(MPC-004) | Low Dose Colchicine(MPC-004) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/74 | 0/59
Other Adverse Events (participants affected / at risk) | 40/52 | 27/74 | 16/59
OTHER ADVERSE EVENTS (reported when occurring in more than 1.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Colchicine(MPC-004) (N=52) | Low Dose Colchicine(MPC-004) (N=74) | Placebo (N=59)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 40 (41) | 17 (18) | 8 (8)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 3 (3)
Vomiting (General disorders) | 9 (9) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotrasnferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glucose Urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein Urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Phosphorous Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urinary Casts (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days